CLINICAL TRIAL: NCT01439568
Title: A Randomized Phase 2 Study of LY2510924 and Carboplatin/Etoposide Versus Carboplatin/Etoposide in Extensive-Stage Small Cell Lung Carcinoma
Brief Title: A Study of LY2510924 in Participants With Extensive-Stage Small Cell Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14242; I2V-MC-CXAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-06

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma
Keywords: Cancer; Lung; Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — LY2510924; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- LY2510924 + Carboplatin + Etoposide (Experimental): LY2510924: 20 milligram (mg) administered once daily as a subcutaneous(SC) injection on days 1 to 7 of the 21 day cycle; repeat every 21 days for 6 cycles. Carboplatin: 5 milligram/millimeter/per minute (mg/mL/min) area under the curve (AUC) administered intravenously on day 1 of the 21 day cycle; repeat every 21 days for 6 cycles.
  Etoposide: 100 milligram square meter (mg/m^2) administered intravenously on days 1 to 3 of the 21 day cycle; repeat every 21 days for 6 cycles.
  Interventions: Drug: LY2510924; Drug: Carboplatin; Drug: Etoposide
- Carboplatin + Etoposide (Active Comparator): Carboplatin: 5 mg/mL/min area under the curve administered intravenously on day 1 of the 21 day cycle; repeat every 21 days for 6 cycles.
  Etoposide: 100 milligram square meter (mg/m^2) administered on days 1 to 3 of the 21 day cycle; repeat every 21 days for 6 cycles.
  Interventions: Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: LY2510924 — Administered subcutaneous injection
  Arms: LY2510924 + Carboplatin + Etoposide
Drug: Carboplatin — Administered intravenously
Drug: Etoposide — Administered intravenously

SUMMARY:
The purpose of this trial is to compare the progression free survival of LY2510924 + carboplatin + etoposide therapy versus carboplatin + etoposide therapy in participants with extensive-stage disease small cell lung cancer (SCLC)

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed extensive-stage disease small cell lung carcinoma
* measurable disease as defined by the New Response Evaluation Criteria in Solid Tumors (RECIST): Revised RECIST Guideline (version 1.1)
* no prior systemic chemotherapy, immunotherapy, biological, hormonal, or investigational therapy for SCLC
* a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale
* adequate organ function, including:

  * hematologic: absolute neutrophil (segmented and bands) count (ANC) greater than or equal to (≥)1.5 x 10^9/ liter (L), platelets ≥100 x 10^9/L, and hemoglobin ≥9 grams per deciliter (g/dL).
  * hepatic: bilirubin less than or equal to (≤)1.5 times upper limits of normal (ULN), and alkaline phosphatase (AP), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 times ULN (AP, AST, and ALT ≤5 times ULN is acceptable if liver has tumor involvement
  * renal: calculated creatinine clearance (CrCl) ≥45 milliliters per minute (mL/min) based on the standard Cockcroft and Gault formula
* For women: Must be surgically sterile (surgical procedure: bilateral tubal ligation), post-menopausal (at least 12 consecutive months of amenorrhea), or compliant with a medically approved contraceptive regimen (intrauterine device [IUD], birth control pills, or barrier device) during and for 6 months after the treatment period; must have a negative serum or urine pregnancy test within 7 days before study enrollment, and must not be breast-feeding. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 6 months after the treatment period.
* estimated life expectancy of at least 12 weeks
* written informed consent prior to any study-specific procedures
* able and willing to learn to self-administer LY2510924, or have a caregiver who is willing to learn and able to administer LY2510924 by subcutaneous (SC) injection

Exclusion Criteria:

* currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* prior treatment with carboplatin/etoposide or LY2510924
* any concurrent administration of any other antitumor therapy
* diagnosis of non-small cell lung cancer (NSCLC) or mixed NSCLC and small cell lung cancer (SCLC)
* no prior malignancy other than SCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated 5 or more years prior to study entry with no subsequent evidence of recurrence. Participants with a history of low grade (Gleason score ≤6) localized prostate cancer will be eligible even if diagnosed less than 5 years prior to study entry
* serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the participant's ability to adhere to the study requirements
* active or ongoing infection during screening requiring the use of systemic antibiotics
* serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease as defined by the New York Heart Association Class III or IV
* clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously- treated central nervous system (CNS) metastases, are asymptomatic, and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug.
* known or suspected allergy to any agent given in association with this trial
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pensacola, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Ventz S, Khozin S, Louv B, Sands J, Wen PY, Rahman R, Comment L, Alexander BM, Trippa L. The design and evaluation of hybrid controlled trials that leverage external data and randomization. Nat Commun. 2022 Oct 2;13(1):5783. doi: 10.1038/s41467-022-33192-1. PMID 36184621
- [Derived] Salgia R, Stille JR, Weaver RW, McCleod M, Hamid O, Polzer J, Roberson S, Flynt A, Spigel DR. A randomized phase II study of LY2510924 and carboplatin/etoposide versus carboplatin/etoposide in extensive-disease small cell lung cancer. Lung Cancer. 2017 Mar;105:7-13. doi: 10.1016/j.lungcan.2016.12.020. Epub 2016 Dec 31. PMID 28236984

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died (any cause) or had disease progression were considered to be study completers.
Groups:
- LY2510924 + Carboplatin + Etoposide: LY2510924: 20 milligram (mg) administered once daily as a subcutaneous injection on days 1 to 7 of the 21 day cycle; repeat every 21 days for 6 cycles. Carboplatin: 5 milligram/millimeter/per minute (mg/mL/min) area under the curve (AUC) administered intravenously on day 1 of the 21 day cycle; repeat every 21 days for 6 cycles. Etoposide: 100 milligram square meter (mg/m^2) administered intravenously on days 1 to 3 of the 21 day cycle; repeat every 21 days for 6 cycles.
Period: Overall Study
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide
Started | 47 | 43
Received at Least One Dose of Study Drug | 47 | 43
Completed | 44 | 41
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide | Total
Number analyzed (Participants) | 47 | 43 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.69 (9.033) | 67.07 (8.328) | 65.31 (8.820)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 22 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 45 | 40 | 85
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 43 | 40 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 43 | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the first date of objectively determined progressive disease (PD) or death from any cause. For participants who are still alive at the time of analysis and without evidence of tumor progression, PFS will be censored at the date of the most recent objective progression-free observation. For participants who receive subsequent anticancer therapy (except PCI) prior to objective disease progression or death, PFS will be censored at the date of the last objective progression-free observation prior to the date of subsequent therapy.
Time Frame: Randomization to Measured Progressive Disease or Date of Death from Any Cause (Up To 59 Months)
Population: All participants who received at least one dose of study drug. One participant was excluded from analysis due to protocol violation.The number of participants censored were LY2510924 + Carboplatin + Etoposide=13 and Carboplatin + Etoposide=7.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide
Number analyzed (Participants) | 47 | 42
Months | 5.88 [4.83 to 6.24] | 5.85 [4.63 to 6.51]
Statistical Analysis 1: Comparison: LY2510924 + Carboplatin + Etoposide vs Carboplatin + Etoposide; Test type: Superiority; p = 0.8072, Logrank Test; Hazard Ratio (HR) = 1.0608, 95% CI 2-sided [0.6598 to 1.7055]

2. Secondary Outcome: Number of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate[ORR])
Description: ORR is defined as the number of participants with a best response of CR and PR defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.Tumor marker results must have normalized. PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD)is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of one or more new lesions is also considered progression.
Time Frame: Baseline to Date of Tumor Response or Measured Progressive Disease or Date of Death from any Cause (Up to 59 Months)
Population: All participants who received at least one dose of study drug. One participant was excluded from analysis due to protocol violation.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide
Number analyzed (Participants) | 47 | 42
Participants | 35 | 34

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the randomization to the date of death from any cause. For participants who are still alive as of the data cutoff date, OS time will be censored on the date of the participant's last contact (last contact for participants in postdiscontinuation is last known alive date in mortality status).
Time Frame: Randomization to Date of Death from Any Cause (Up To 59 Months)
Population: All participants who received at least one dose of study drug. One participant was excluded from analysis due to protocol violation. The numbers of participants censored were LY2510924 + Carboplatin + Etoposide= 4 and Carboplatin + Etoposide=3.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide
Number analyzed (Participants) | 47 | 42
Months | 9.72 [6.64 to 11.70] | 11.14 [8.25 to 14.23]

4. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Tumor marker results must have normalized. PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD)is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Date of Response to Date of Progressive Disease (Up To 59 Months)
Population: All participants who received at least one dose of study drug. One participant was excluded from analysis due to protocol violation. The number of participants censored were LY2510924 + Carboplatin + Etoposide=47 and Carboplatin + Etoposide=42.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide
Number analyzed (Participants) | 47 | 42
Months | 4.83 [3.58 to 5.09] | 4.67 [3.32 to 5.78]

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | LY2510924 + Carboplatin + Etoposide | Carboplatin + Etoposide
Serious Adverse Events (participants affected / at risk) | 24/47 | 13/43
Other Adverse Events (participants affected / at risk) | 47/47 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2510924 + Carboplatin + Etoposide (N=47) | Carboplatin + Etoposide (N=43)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2510924 + Carboplatin + Etoposide (N=47) | Carboplatin + Etoposide (N=43)
Anaemia (Blood and lymphatic system disorders) | 28 (94) | 21 (81)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 13 (18) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 28 (43) | 22 (49)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (56) | 17 (52)
Tachycardia (Cardiac disorders) | 3 (4) | 2 (2)
Vision blurred (Eye disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 18 (20) | 18 (22)
Diarrhoea (Gastrointestinal disorders) | 12 (16) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 5 (10) | 3 (4)
Nausea (Gastrointestinal disorders) | 23 (44) | 19 (36)
Vomiting (Gastrointestinal disorders) | 15 (21) | 8 (10)
Asthenia (General disorders) | 6 (7) | 6 (7)
Chest pain (General disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 29 (46) | 25 (46)
Injection site erythema (General disorders) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 9 (11) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 7 (11) | 10 (10)
Pain (General disorders) | 5 (5) | 4 (5)
Pyrexia (General disorders) | 5 (9) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (5) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 3 (3)
Blood magnesium decreased (Investigations) | 3 (3) | 1 (1)
Blood uric acid increased (Investigations) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (6) | 3 (6)
Neutrophil count increased (Investigations) | 3 (6) | 1 (2)
Platelet count decreased (Investigations) | 3 (7) | 3 (6)
Weight decreased (Investigations) | 6 (6) | 6 (7)
White blood cell count increased (Investigations) | 5 (9) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 13 (15) | 11 (13)
Dehydration (Metabolism and nutrition disorders) | 8 (9) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (11) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (12) | 7 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 7 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (12) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (4)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (7) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 8 (8)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (5)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 11 (12) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 12 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 10 (13)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (27) | 17 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (4)
Flushing (Vascular disorders) | 4 (5) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days